CLINICAL TRIAL: NCT02422225
Title: Improvement of Swallowing Function of Stroke Patients by Dual Transcranial Direct Current Stimulation(tDCS)
Brief Title: A Study of tDCS for Swallowing Difficulties in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Associate Professor, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNUYH-03-2015-004
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eldith DC-STIMULATOR group (Experimental): Intervention:
  20-minutes of transcranial Direct Current Stimulation (tDCS) application 5 days a week for 2 weeks (30 applications for each 3 groups: total 90 applications)
  Interventions: Device: Eldith DC-STIMULATOR
- sham-Eldith DC-STIMULATOR group (Sham Comparator): Intervention: 20-minutes of sham-tDCS application 5 days a week for 2 weeks (total 30 applications)
  Interventions: Device: Sham Eldith DC-STIMULATOR

INTERVENTIONS:
Device: Eldith DC-STIMULATOR — Transcranical direct current stimulator (Neuroconn GmbH, Ilmenau, Germany) approved by Conformity European as safe treatment device for stroke patients
  tDCS intervention]
  * Intensity: 1.5mA for 20min Device: Neuroconn GmbH, Ilmenau, Germany
  * Stimulation site <Experimental group>
    * Anode-Anode dual stimulation group Anode: affected pharyngeal motor cortex / Cathode: affected supraorbit Anode: non-affected pharyngeal motor cortex / Cathode: non-affected supraorbit
    * Anode-Cathode dual stimulation group Anode: affected pharyngeal motor cortex Cathode: non-affected pharyngeal motor cortex
    * Single stimulation group Anode: affected pharyngeal motor cortex Cathode: non-affected supraorbit <Control group> Sham stimulation
  Arms: Eldith DC-STIMULATOR group
Device: Sham Eldith DC-STIMULATOR
  Arms: sham-Eldith DC-STIMULATOR group

SUMMARY:
The primary objective of this study is to investigate whether the dual transcranial direct current stimulation(tDCS) improves the swallowing function of stroke patients.

DETAILED DESCRIPTION:
120 patients were recruited and randomized to receive either real or sham-tDCS. Real experimental groups were divided into three types; Anode-Anode dual stimulation group, Anode-Cathode dual stimulation group, Single stimulation group. 20-minutes session of the stimulation were applied 5 times a weeks for 2 weeks at pharyngeal motor cortex of affected or non-affected site. The patients were evaluated at baseline, immediately and 2 weeks after tDCS.

ELIGIBILITY:
Inclusion Criteria

* Subjects who have diagnosed as primary stroke by physician's physical exam or radiologic diagnosis
* Subjects who have cortical or subcortical brain lesion
* Subjects who was diagnosed as stroke within 6 months
* Subjects ages from 18years to 80years old
* Subjects who have less than 5 points of DOSS score due to swallowing difficulty from CNS injury
* Subjects who is possible to receive swallowing function intervention 5 days a week
* Subjects who understand the purpose of the study and acquired the consent of the patient or caregiver
* Subjects who had no effect from brain stimulation or electrical stimulation therapy

Exclusion Criteria

* Subjects who have pre-existing and active major neurological disease
* Subjects who have pre-existing and active major psychiatric disease, such as major depression, schizophrenia, bipolar disease, or dementia
* Subjects who have brain lesion except cortex or subcortex area
* Subjects who have any metal component after brain surgery, low threshold to pain, history of seizure
* Subjects who is estimated as not appropriate for the study by the investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Dysphagia Outcome and Severity Scale(DOSS) from video fluoroscopic swallowing study(VFSS) | up to 60 sec

SECONDARY OUTCOMES:
American Speech-LanguageHearing Association(ASHA)-Norms | up to 2 weeks after tDCS
  Change in swallowing function
Korean Version of Modified Barthel Index(K-MBI) | up to 2 weeks after tDCS
  Change in activity of daily living
Dysphagia Outcome and Severity Scale(DOSS) from video fluoroscopic swallowing | 2 weeks after tDCS
  Change in swallowing function

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Il Shin, Ph.D., Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

REFERENCES:
- [Background] Lequerica AH, Kortte K. Therapeutic engagement: a proposed model of engagement in medical rehabilitation. Am J Phys Med Rehabil. 2010 May;89(5):415-22. doi: 10.1097/PHM.0b013e3181d8ceb2. PMID 20407308